CLINICAL TRIAL: NCT01289041
Title: A Phase II, Single-arm Study of Orally Administered BKM120 as Second-line Therapy in Patients With Advanced Endometrial Carcinoma
Brief Title: BKM120 as Second-line Therapy for Advanced Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120C2201; 2010-022015-19 (EudraCT Number)
Record Dates: First submitted 2011-01-26; First posted 2011-02-03 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Advanced Endometrial Cancer
Keywords: Advanced endometrial cancer; PI3K pathway; second-line treatment
MeSH Terms: interventions — NVP-BKM120

ARMS (1):
- All Patients (Experimental)
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120
  Other Names: Buparlisib

SUMMARY:
This is a prospective multi-center, open-label, single arm, Phase II study to investigate the safety and efficacy of BKM120 in patients with advanced endometrial carcinoma whose disease progressed on or after a first-line antineoplastic treatment. Patients will receive BKM120 orally at a dose of 100 mg/day. Availability of tumor specimen (either archival tissue or a fixed fresh biopsy) is mandatory for assessment of the PI3K (Phosphatidylinositol 3 Kinase (PI3K) pathway activation status.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2
* histologically confirmed diagnosis of advanced endometrial carcinoma with available tissue specimen for identification of PI3K pathway activation (archival tissue or a fixed fresh biopsy)
* one prior line of antineoplastic treatment with a cytotoxic agent
* objective progression of disease after prior treatment and at least one measurable lesion as per RECIST criteria
* adequate bone marrow and organ function

Exclusion Criteria:

* previous treatment with PI3K and/or mTOR inhibitors
* symptomatic CNS metastases
* concurrent malignancy or malignancy within 3 years of study enrollment
* Active mood disorder as judged by investigator or medically documented history of mood disorder (e.g. major depressive episode, bipolar disorder, obsessive-compulsive disorder, schizophrenia, etc.), ≥ CTCAE grade 3 anxiety
* pelvic and/or para-aortic radiotherapy ≤ 28 days prior to enrollment in the study
* poorly controlled diabetes mellitus (HbA1c > 8 %)
* history of cardiac dysfunction or active cardiac disease as specified in the protocol
* impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (39):
- United States (9):
  - St. Joseph's Hospital & Medical Center St Joseph's, Phoenix, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Morristown Memorial Hospital MMH, Morristown, New Jersey
  - Carolinas HealthCare Systems Blumenthal Cancer Center, Charlotte, North Carolina
  - University of Oklahoma Health Sciences Center OU Health, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute SCRI (2), Nashville, Tennessee
  - Texas Oncology, P.A. Austin, Bedford, Texas
  - South Texas Oncology and Hematology, PA South Tex Onc, San Antonio, Texas
  - Cancer Care Northwest CC Northwest- Spokane South(3), Spokane, Washington
- Novartis Investigative Site, Parkville, Victoria, Australia
- Belgium (3):
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (4):
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Mainz
- Italy (5):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Napoli
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Singapore, Singapore
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 70
Completed | 0
Not Completed | 70
Not completed — Adverse Event | 24
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 41
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.04)
Sex/Gender, Customized [Number; unit: participants]
  Female | 70
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (BORR) According to PI3K Activation Pathway Status
Description: BOR was determined based on investigator assessment of overall lesion response using RECIST criteria guidelines. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 24 months
Population: Full analysis set includes all patients who received at least one dose of study drug.
Measure: Number; unit: number of participants
Arm/Group | Activated Pl3K | Non-Activated Pl3K | All Patients
Number analyzed (Participants) | 49 | 21 | 70
number of participants
  Patients with Measurable disease at baseline | 49 | 21 | 70
  Complete Response (CR) | 1 | 0 | 1
  Partial Response (PR) | 0 | 1 | 1
  Stable Disease (SD) | 19 | 7 | 26
  Progressive disease (PD) | 20 | 9 | 29
  Unknown (UNK) | 9 | 4 | 13
  Overall Response Rate (CR + PR) | 1 | 1 | 2

2. Secondary Outcome: Progression Free Survival (PFS) According to PI3K Activation Pathway Status
Description: PFS is defined as the time from start of treatment to the date of first documented progression or death due to any cause. If a patient has not had an event, PFS will be censored at the date of last adequate tumor assessment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 months
Population: Full analysis set includes all patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Activated Pl3K | Non-Activated Pl3K | All Patients
Number analyzed (Participants) | 49 | 21 | 70
months | 1.9 [1.8 to 3.2] | 1.9 [1.6 to 3.3] | 1.9 [1.8 to 2.8]

3. Secondary Outcome: Overall Survival (OS) According to PI3K Activation Pathway Status
Description: Overall survival (OS) was defined as the time from start of treatment to the date of death due to any cause. If a patient is not known to have died, survival was censored at the last date of contact. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
Population: Full analysis set includes all patients who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Activated Pl3K | Non-Activated Pl3K | All Patients
Number analyzed (Participants) | 49 | 21 | 70
months | 8.9 [6.3 to 16.2] | 14.2 [8.6 to 24.0] | 9.9 [7.4 to 16.2]

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 33/70
Other Adverse Events (participants affected / at risk) | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=70)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Erosive oesophagitis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Face oedema (General disorders) | 1
Hypersensitivity (Immune system disorders) | 3
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Uterine infection (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
International normalised ratio increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hypercreatininaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=70)
Anaemia (Blood and lymphatic system disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 9
Dysphagia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 31
Stomatitis (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 14
Asthenia (General disorders) | 6
Fatigue (General disorders) | 24
Oedema peripheral (General disorders) | 9
Pain (General disorders) | 4
Pyrexia (General disorders) | 6
Urinary tract infection (Infections and infestations) | 10
Alanine aminotransferase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 18
Blood alkaline phosphatase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 11
Weight decreased (Investigations) | 14
Decreased appetite (Metabolism and nutrition disorders) | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 37
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 10
Headache (Nervous system disorders) | 8
Memory impairment (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 17
Confusional state (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 16
Insomnia (Psychiatric disorders) | 8
Mood altered (Psychiatric disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 21
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial